CLINICAL TRIAL: NCT04315142
Title: Transcutaneous Tibial Nerve Stimulation (TTNS) for Treating Neurogenic Lower Urinary Tract Dysfunction: A Multicentre, Randomised, Sham-controlled, Double-blind Clinical Trial
Brief Title: Bladder and TranscUtaneous Tibial Nerve Stimulation for nEurogenic Lower Urinary Tract Dysfunction
Acronym: bTUNED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting participants
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: bTUNED
Record Dates: First submitted 2020-03-09; First posted 2020-03-19 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-11

CONDITIONS: Neurogenic Bladder Dysfunction
Keywords: Randomized; Sham-controlled; Transcutaneous tibial nerve stimulation (TTNS); Neurogenic detrusor overactivity; Neuromodulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcutaneous tibial nerve stimulation (TTNS) (Experimental)
  Interventions: Device: Experimental TTNS
- TTNS sham stimulation (Sham Comparator)
  Interventions: Device: Sham TTNS

INTERVENTIONS:
Device: Experimental TTNS — 30-minute TTNS intervention is performed 2 days a week during a treatment period of 6 weeks
  Arms: Transcutaneous tibial nerve stimulation (TTNS)
Device: Sham TTNS — 30-minute sham intervention is performed 2 days a week during a treatment period of 6 weeks
  Arms: TTNS sham stimulation

SUMMARY:
Many patients with neurological diseases suffer from neurogenic lower urinary tract dysfunction (NLUTD), which often severely impairs quality of life, due to urinary urgency with or without incontinence and voiding dysfunction. In addition, the upper urinary tract may be jeopardized because of high intravesical pressure caused by detrusor overactivity (DO) with concurrent detrusor-sphincter-dyssynergia and/or low bladder compliance.

The treatment of NLUTD is a challenge since conventional conservative therapies often fail and more invasive treatments such as intradetrusor onabotulinumtoxinA injections, bladder augmentation and urinary diversion have to be considered. Neuromodulation therapies including tibial nerve stimulation (TNS) may be alternative non-invasive treatment options.

Indeed, TNS is an effective and safe treatment for idiopathic overactive bladder proven in randomised controlled trials (RCTs), but its value in neurological patients is unclear. In a recent systematic review, the investigators found evidence that TNS might become a promising treatment option for NLUTD, however, more reliable data from well-designed RCTs are urgently needed to reach definitive conclusions.

However, this study will be the first adequately sampled and powered, randomised, sham-controlled, double-blind trial assessing transcutaneous TNS (TTNS) for NLUTD. It will provide significant insights into the efficacy of TTNS in patients suffering from NLUTD and in the case that this treatment is really effective in the neurological population, the investigators findings would completely revolutionize the management of NLUTD in daily clinical practice. Moreover, this interdisciplinary clinical trial will relevantly influence the neurological and urological approach in the management of NLUTD promoting future collaborative projects improving patients' medical care and underlying the pioneering role of Switzerland in the rapidly developing and ambitious research field of neuro-urology.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age ≥18 years
* Last urethro-cystoscopy and bladder washing cytology within 1 year before inclusion
* Last urodynamic investigation within 6 months and no change of bladder medication since then
* Refractory LUTD due to a neurological disorder:

  1. Neurogenic OAB (i.e. urgency frequency syndrome with or without urgency incontinence) refractory to antimuscarinics (pharmacotherapy for at least 4 weeks with at least 2 antimuscarinics)
  2. Neurogenic voiding dysfunction (i.e. incomplete bladder emptying/incomplete / complete urinary retention) refractory to alpha-blocker (pharmacotherapy with an alpha-blocker for at least 4 weeks)
  3. Combination of neurogenic OAB and neurogenic voiding dysfunction (i.e. urgency frequency syndrome with or without urgency incontinence and incomplete / complete urinary retention) refractory to antimuscarinics (pharmacotherapy for at least 4 weeks with at least 2 antimuscarinics) and alpha-blocker (pharmacotherapy with an alpha- blocker for at least 4 weeks)
* Motor response induced by TTNS stimulation at least at one leg
* Willing not to change or start any new medications or treatments for the LUT during the entire study period (from screening till unblinding)

Exclusion Criteria:

* Contraindications to the investigational product
* Known or suspected non-adherence, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia
* Participation in another study with investigational drug or product within the 30 days preceding and during the present study
* Neuromodulation treatment for urological indication in the last six months or ongoing
* Botulinum toxin injections in the detrusor and/or urethral sphincter in the last six months
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Individuals especially in need of protection (according to Research with Human Subjects published by the Swiss Academy of Medical Sciences [www.samw.ch/en/News/News.html]
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Success of TTNS | study week 8 / study end
  Success of TTNS defined as:
  * ≥50% reduction in incontinence rates per 24 hours and/or ≥50% reduction in micturition/catheterization frequency per 24 hours in patients with neurogenic overactive bladder (OAB)
  * Reduction of post void residual (PVR) below 25% of bladder capacity if bladder capacity
    * 100 mL, or below 50% of bladder capacity if bladder capacity <100 mL in patients with neurogenic voiding dysfunction
  * In patients with combined neurogenic OAB and neurogenic voiding dysfunction: The success criteria of leading symptom/dysfunction will be chosen

SECONDARY OUTCOMES:
Volumetric changes during urodynamics and their relation to clinical outcomes | Baseline; study week 8 / study end
  Cystometric capacity [mL], volume at first DO [mL], voided volume [mL] and post void residual [mL] as assessed by urodynamic measurement
Changes in bladder compliance [mL/cmH2O] during urodynamics and their relation to clinical outcomes | Baseline; study week 8 / study end
Pressure changes during urodynamics and their relation to clinical outcomes | Baseline; study week 1-8 / study end
  Maximum DO pressure [cmH2O], detrusor leak-point pressure [cmH2O], maximum detrusor pressure [cmH2O] during storage phase, maximum detrusor pressure [cmH2O] during voiding phase, detrusor pressure at maximum flow rate [cmH2O] as assessed by urodynamic measurement
Changes in maximum flow rate [mL/s] as assessed by urodynamics and their relation to clinical outcomes | Baseline; study week 8 / study end
Changes in vesicoureterorenal reflux (VUR) as assessed by videography during urodynamics and their relation to clinical outcomes | Baseline; study week 8 / study end
Changes in pelvic floor activity as assessed by electromyography (EMG) during urodynamics and their relation to clinical outcomes | Baseline; study week 8 / study end
Changes in bladder storage and voiding parameters and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; study week 8 / study end
  Assessed by a bladder diary
Changes in bowel diary parameters and their relation to clinical outcomes | Baseline; study week 8 / study end
  Assessed by a bowel diary
Goal attainment scaling assessed by a self-assessment goal achievement (SAGA) questionnaire | Baseline; study week 8 / study end
  The baseline SAGA module asks patients to rate the importance of 9 prespecified (fixed) treatment goals that describe reducing the following LUTS: frequency (daytime and nighttime); sensation of pressure; primary sensation to use the bathroom; bladder voiding; starting or maintaining a urine stream; urine loss when coughing, laughing, exercising, or sneezing; urine leakage; and urgency. In addition to the 9 fixed goals, patients can list up to 5 additional (open) treatment goals. Patients rate the importance of each goal using a 5-point scale ranging from "not very important goal" to "very important goal." In the SAGA follow-up module, patients rate their achievement of each individualized goal and overall goal achievement with a 5-point scale ranging from "did not achieve goal" to "greatly exceeded goal."
Changes in International Prostate Symptom (IPSS) questionnaire and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; study week 8 / study end
  The IPSS ("International Prostate Symptom Questionnaire") score is based on questions concerning urinary symptoms and quality of life (QoL). It consists of 8 items covering 7 urinary symptoms related dimensions (subscales) and 1 additional item assessing quality of life. Each item is rated on a 6-point scale (0=not at all; 5=almost always). The lowest possible score in the total IPSS score is 0 (asymptomatic); the highest possible score is 35 (symptomatic). The QoL index is rated on a 7-point scale, with 0 indicating "delighted" and 6 "terrible."
Changes in urinary symptoms as assessed by the Urinary Symptom Profile (USP) questionnaire and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; study week 8 / study end
  The USP ("Urinary Symptom Profile") score is based on questions concerning urinary symptoms and their severity in males and females. It consists of 13 items covering 3 dimensions (subscales) with 7 overactive bladder (OAB), 3 stress urinary incontinence (SUI), and 3 low stream (LS) related items. Each item is rated on a 4-point scale. The lowest score is 0 (asymptomatic); the highest score is 3 (symptomatic).
Changes in Qualiveen questionnaire scores and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; study week 8 / study end
  Qualiveen-30 assesses the Specific Impact of Urinary Problems (SIUP) on Quality of Life. It consists of 30 items covering 4 domains, namely inconvenience (9 questions), restrictions (8 questions), fears (8 questions), and impact on daily life (5 questions). Each item is rated on a 5-point ordinal scale (0=asymptomatic; 4=symptomatic). The index of the SIUP on Quality of Life is the mean of the four individual scores. The lowest possible overall score in the Qualiveen-30 is 0 (Urinary problems have no specific impact on QoL); the highest possible score is 30 (Urinary problems have a huge specific impact on QoL).
Changes in Female Sexual Function Index (FSFI) and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; study week 8 / study end
  The FSFI ("Female Sexual Function Index") is based on questions concerning female sexual functions. It consists of 19 items covering 6 domains, namely sexual desire, arousal (both subjective and physiologic), lubrication, orgasm, satisfaction, and pain. The lowest possible score in the total FSFI is 2 (asymptomatic); the highest possible score is 36 (symptomatic).
Changes in International Index of Erectile Function (IIEF) and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; study week 8 / study end
  The IIEF ("International Index of Erectile Function") is based on questions concerning erectile dysfunction. It consists of 15 items covering 5 domains, namely erectile functioning, orgasmic functioning, sexual desire, and intercourse satisfaction along with a fifth component which encompasses the concept of overall sexual satisfaction. While items 1-10 are rated on a 6-point Likert-type scale from 0 to 5, items 11-15 are rated on a 5-point Likert-type scale from 1 to 5. Higher scores are reflecting less dysfunction. Domain scores are computed by summing the sores for individual items in each domain.
Variability and validity of University of South Australia Urinary Symptom Assessment questionnaire (USA2) for treatment follow-up | Baseline; once per week during the TTNS intervention period; study week 8 / study end
  The USA2 ("University of South Australia Urinary Symptom Assessment") assesses multiple dimensions of urgency sensation. 10 items are rated on a 6-point Likert-type scale from 0 to 5. Lower scores are reflecting lesser urgency symptoms. Domain scores are computed by summing the sores for individual items in each domain.
Changes in Neurogenic Bowel Dysfunction (NBD) questionnaire and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; study week 8 / study end
  The NBD ("Neurogenic Bowel Dysfunction") score is based on questions concerning constipation and fecal incontinence and was developed for and validated in the spinal cord injury population. It consists of 10 items. The lowest possible score in the total NBD is 0 (asymptomatic); the highest possible score is 47 (symptomatic). The interpretation of the total NBD score is very minor NBD (0-6), minor NBD (7-9), moderate NBD (10-13), and severe NBD (≥14).
Changes in neurophysiology measurements of evoked potentials (EPs) as well as nerve conduction measurements and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; study week 8 / study end
Volumetric changes during rectal sensitivity testing and barostat assessment and their relation to clinical outcomes | Baseline; study week 8 / study end
  Initial sensation [mL], volume at urge to defecate [mL], maximum tolerated volume [mL] as assessed by rectal sensitivity testing; rectal capacity [mL] assessed by barostat assessment
Pressure changes during anorectal manometry and barostat assessment and their relation to clinical outcomes | Baseline; study week 8 / study end
  Basal Internal anal sphincter pressure [mmHg], squeeze external anal sphincter pressure [mmHg], relaxation internal anal sphincter pressure during defecation [mmHg], intraabdominal pressure during defecation [mmHg]
Changes in rectal compliance [mL/cmH2O] during anorectal manometry and barostat assessment and their relation to clinical outcomes | Baseline; study week 8 / study end
Changes in defecatory disorder [Rao's classification] identified during anorectal manometry and their relation to clinical outcomes | Baseline; study week 8 / study end
  Anorectal manometry is the preferable test for defecatory disorder. Rao's classification describes the four types manometric patterns (I-IV) that are identified through manometric assessments.
Incidence of side effects as well as number and intensity/severity (mild/moderate/severe) of AEs and SAE | During complete study period
  Categories:
  * infection - Urinary Tract Infection (UTI)
  * infection - other than UTI
  * skin irritation at the electrode site
  * pressure ulcer
  * severe neurological deterioration
  * severe or sudden increase in pain
  * severe or sudden increase in spasticity
  * deep vein thrombosis / pulmonary embolism
  * autonomic dysreflexia
  * urgent (unexpected) transfer/admittance to an acute care facility

CONTACTS AND LOCATIONS:
Locations (12):
- University Hospital Antwerp, Edegem, Belgium
- University of Sao Paulo School of Medicine, São Paulo, Brazil
- Italy (2):
  - Careggi University Hospital, Florence
  - Tor Vergata University Hospital, Rome
- Switzerland (8):
  - Inselspital Bern, University Hospital, Bern, Canton of Bern
  - Cantonal Hospital Winterthur, Winterthur, Canton of Zurich
  - Cantonal Hospital Aarau, Aarau
  - REHAB Basel, Basel
  - EOC - Regional Hospital Bellinzona and Valleys, Bellinzona
  - Centre hospitalier universitaire vaudois CHUV, Lausanne
  - Cantonal Hospital St. Gallen, Sankt Gallen
  - Balgrist University Hospital, Zurich

REFERENCES:
- [Derived] Stalder SA, Gross O, Anderson CE, Bachmann LM, Baumann S, Birkhauser V, Bywater M, Del Popolo G, Engeler DS, Agro EF, Friedl S, Grilo N, Kiss S, Koschorke M, Leitner L, Liechti MD, Mehnert U, Musco S, Sadri H, Stachele L, Tornic J, van der Lely S, Wyler S, Kessler TM. bTUNED: transcutaneous tibial nerve stimulation for neurogenic lower urinary tract dysfunction. BJU Int. 2023 Sep;132(3):343-352. doi: 10.1111/bju.16081. Epub 2023 Jun 13. PMID 37204144